CLINICAL TRIAL: NCT01328990
Title: Pharmacokinetics of Sulfadoxine-pyrimethamine Plus Amodiaquine When Used for Malaria Intermittent Preventive Treatment in Children
Brief Title: Pharmacokinetics of Sulfadoxine-pyrimethamine Plus Amodiaquine for Intermittent Preventive Treatment in Children (IPTc)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Cheikh Anta Diop University, Senegal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IZ5856
Record Dates: First submitted 2011-04-04; First posted 2011-04-05 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Malaria
Keywords: IPTc; malaria; children; pharmacokinetics; amodiaquiane; sulfadoxine-pyrimethamine
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine plus amodiaquine — one dose of sulfadoxine-pyrimethamine 25/1.25 mg/kg plus three daily doses of amodiaquine, 10 mg/kg/day

SUMMARY:
The aim of the study is to determine the pharmacokinetic profile of sulfadoxine-pyrimethamine plus amodiaquine (SP+AQ) when used for seasonal Intermittent Preventive Treatment (IPT) to prevent malaria in children aged 3 to 59 months in Lamarame, NDoffane District, Senegal. Several studies have shown that seasonal IPT in children can provide a high degree of protection against clinical malaria. SP+AQ is the most effective regimen. However little is known about the pharmacokinetics of amodiaquine and sulfadoxine-pyrimethamine in children. The purpose of this study is to determine the pharmacokinetics profile of SP+AQ when used for IPT in Senegalese children. 150 children aged 3 to 59 months will be enrolled in November. They will receive a therapeutic dose of sulfadoxine-pyrimethamine and amodiaquine, and will be followed up for 30 days. Four finger prick blood samples will be taken from each child for PK analysis.

DETAILED DESCRIPTION:
SP+AQ is the most effective regimen for IPT in children, but there is little information about the pharmacokinetics of these drugs in children. Although this combination has been used for many years for treatment of clinical malaria there have been no studies of the pharmacokinetics of this combination. A recent study described the pharmacokinetics of amodiaquine when used in combination with artesunate to treat children with clinical malaria (Stepniewska et al, 2009), and another recent study described the pharmacokinetics of SP in children with malaria (Barnes et al, 2006), and a further study of SP in children with uncomplicated malaria demonstrated a low plasma level of the drug in children who failed the treatment (Obua et al. 2008), but there are no studies of these drugs given together or in healthy children. This information is important in order to check the bioavailability of the two drugs when used for IPT and to check the adequacy of the currently recommended dosage. The study will be conducted in a rural district of Senegal, after holding community meetings to explain the study. 150 children aged 1-5 years, boys and girls who do not have history of allergy to study drugs and whose parents agreed for them to participate will be enrolled at the study clinic. The sample size determination is based on experience from other PK studies. During the study organization phase, meetings will be held at the health facilities, members of the community, community leaders, and health staff will be invited to attend, the investigators will explain, in local language, the aims of the study, the recruitment and follow up procedures, the total sample size needed, and the duration of follow up. The detailed schedule for blood sampling will be explained. Subsequently the investigators will visit families at home to explain the study and invite people to attend at the clinic. Mothers or carers will be asked to bring the child to the clinic where, after signing to indicate consent, the child will be weighed and have a clinical examination, a finger prick blood sample will be taken by drawing blood into a vacutainer, from which 70µL of blood will be pipetted onto filter paper. SP and the first dose of AQ will be administered according to the child's weight, the child will be kept under observation for 30 minutes before being allowed to return home. The remaining doses of amodiaquine (days 1 and 2) will be given to a field worker who will visit the child at home to supervise drug administration. The exact time of the administration will be recorded. Any child who vomits a dose will be given a repeat dose. The child will be asked to provide a finger prick blood sample on three further occasions between day 1 and day 28, determined according to a schedule chosen to allow good estimation of PK parameters. Trained field staff will visit each child on day 4, to ask about any adverse reactions to the drugs, and on day 14 and 28 to check the child is well. Children with signs of severe malaria, or any other severe illness, will be referred immediately to the health post. For other children, if the child has axillary temp >=37.5oC or a history of fever in the last 48 hours a finger prick blood sample will be taken for malaria diagnosis by rapid test and blood film to be read later. Children with a positive test will be treated with Coartem.

ELIGIBILITY:
Inclusion Criteria:

* age 3 months to 5 years
* no allergy to study drugs
* consent from parent or guardian

Exclusion Criteria:

* chronic illness

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Concentration of sulfadoxine, pyrimethamine, and desethylamodiaquine | 28 days
  Concentration of the drugs will be measured at four time points.

SECONDARY OUTCOMES:
Tolerability | 28 days
  Adverse events will be recorded during home visits

CONTACTS AND LOCATIONS:
Overall Officials: Badara Cisse, PhD, Study Chair — Universite Chiekh Anta Diop; Paul Milligan, PhD, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- Universite Chiekh Anta Diop, Dakar, Senegal